CLINICAL TRIAL: NCT03347812
Title: Clinical Study on Evaluation of Total Endovascular Aortic Arch Repair
Brief Title: Clinical Study for Evaluating the Safety and Efficacy of Total Endovascular Aortic Arch Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Peking University People's Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Chang Shu, Director of Vascular Surgery Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: D171100002917004
Record Dates: First submitted 2017-11-05; First posted 2017-11-20 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Aortic Dissection; Aortic Arch Aneurysm; Ulcer; Pseudoaneurysm
Keywords: Aortic Arch; Endovascular Treatment; Traditional Open Surgery; Chimney Technique; Fenestration Technique; Branched Stent-grafts Technique
MeSH Terms: conditions — Aortic Dissection; Aneurysm, Aortic Arch; Ulcer; Aneurysm, False | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular Aortic Repair: Patients with aortic arch lesions who only received endovascular treatment, including chimney / fenestration / branch stent-grafts technique and combination of these techniques, would be assigned to this group.
  Interventions: Procedure: Endovascular Aortic Repair
- Total Arch Replacement: Patients with aortic arch lesions who only received traditional open surgery for total aortic arch replacement, would be assigned to this group.
  Interventions: Procedure: Total Arch Replacement

INTERVENTIONS:
Procedure: Endovascular Aortic Repair — Without surgery to expose the lesion directly, minimal invasive treatment for the aortic arch lesion under the guidance of imaging equipment is performed through the blood vessel with a tiny wound of a few centimeters, in our research, including chimney, branch stent-grafts and fenestration techniques.
  Groups: Endovascular Aortic Repair
Procedure: Total Arch Replacement — A kind of open surgery is performed for the replacement of total aortic arch.
  Groups: Total Arch Replacement

SUMMARY:
Aortic disease is a kind of cardiovascular diseases with very high mortality rate and high risk of surgical treatment. At present, the surgical and endovascular treatment for diseases in the ascending aorta, descending aorta and abdominal aorta are becoming more and more mature. However, due to the complexity of the aortic arch in anatomy, function and pathological changes, the optimal treatment strategy for diseases in the aortic arch has been controversial constantly.

This research is a multi-center(four centers), prospective, controlled, large-scale (about 400 subjects) clinical study, using traditional thoracic surgery of aortic arch disease as a control to verify that new techniques for endovascular treatment is not inferior to traditional thoracic surgery in terms of efficiency and safety.

Further more, the investigators plan to explore the indications of the application of these new techniques, develop a better diagnosis and treatment program, reduce the risk of such surgical treatment and the incidence of complications, improve clinical efficacy and the overall quality of the disease.

DETAILED DESCRIPTION:
The subjects in this study are patients with aortic arch disease, after scientific assessment made by the team with wide experience in aortic open surgery and endovascular treatment, who are able to both withstand traditional total aortic arch replacement (TAR) and are suitable for complete thoracic endovascular aortic repair (cTEVAR) in terms of anatomical structure. According to the requirement of statistical analysis, more than 400 patients would be enrolled in the four centers (Fuwai Hospital, Peking University People's Hospital, China-Japan Friendship Hospital and Beijing Hospital) within 2 years. Combined the actual situation of the patients, subjects would be divided into TAR and cTEVAR groups. During the study, the investigators would collect the data including blood and biochemical indexes, complications, aortic CT examination, surgical procedure, and the follow-up information in discharge, one month after surgery, six months after surgery and twelve months after surgery.

The primary endpoint of this study is one-year treatment success, which means there are no death within 30 days after surgery, no adverse cardiovascular and no cerebrovascular events and no re-operative intervention associated with aorta occurred during the 1-year follow-up period. Secondary endpoints include the occurrence of postoperative leaks, occlusion, stenosis and thrombosis of aortic arch branches, the incidence of device-related adverse events, and the incidence of other serious complications. This study uses the primary endpoint as a measure of efficacy, and the secondary endpoint as a measure of safety for both treatment methods. The primary analysis of collected data would be based on intention-to-treat (ITT) principle, and all enrolled patients would be included in the final analysis.

The Cochran-Mantel-Haenszel (CMH) chi square analysis for adjusting center effects will be used for comparisons of major indicators, estimating differences in success rates and their 95% confidence intervals in two groups. If the lower limit of the 95% Confidence Interval (CI) of the difference in success rate between the test group and control group exceeds the pre-established non-inferiority cutoff, the endovascular treatment can be considered to be as effective as traditional open surgery. The significance level for all statistical tests is 5%, and the statistical analysis software is Statistics Analysis System (SAS) 9.3.

ELIGIBILITY:
Inclusion Criteria:

* Patients have aortic arch lesions caused by atherosclerosis and hypertension, and are also suitable for both chimney/ fenestration / branch stent-grafts technique and total arch replacement surgery simultaneously.
* Lesions involve the aortic arch, at least one branch of the aortic arch to be revascularized.
* The type of lesion is dissection, aneurysm, pseudoaneurysm, or ulcer.
* Life expectancy is more than 1 year.
* Patients are able to understand the purpose of this trial, voluntarily attend and sign the informed consent form, and are willing to accept the specified follow-up at specific time point.

Exclusion Criteria:

* Patients had a stroke or ST-segment elevation myocardial infarction within 30 days prior to surgery.
* Patients underwent major surgery (grade 3 or above) or interventional therapy within 30 days prior to surgery.
* Patients will undergo any major elective surgery (grade 3 or above) or interventional therapy within 30 days after surgery.
* Patients had a previous thoracic aortic surgery in the past.
* Patients had previous thoracic aortic endovascular treatment, and the last implants had an effect on this procedure or had intersections with implants would be used in this procedure.
* Patients need intervention in other vascular lesions (such as coronary arteries, lower extremity arteries, carotid arteries) in the same procedure, or have heart disease and postoperative medication regimens are affected.
* Patients have hepatic and renal insufficiency (serum creatinine> 186umol / L, Child-Pugh grade B, grade C).
* Aortic arch lesions are not caused by atherosclerosis or hypertension, such as connective tissue disease, aortic genetic diseases, etc.
* Aortic arch lesions are caused by Infectious diseases.
* Patients had serious illnesses (eg, severe chronic obstructive pulmonary disease (COPD) , cancer, dementia, etc.), or the physical condition would affect patients' compliance in this study.
* Patients are currently participating in other studies, and the primary endpoint has not been reached.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had aortic arch lesions, need surgery, and are hospitalized in these four hospitals (Fuwai Hospital, Beijing Hospital, China-Japan Friendship Hospital and Peking University People's Hospital) . These four hospitals are all located in Beijing, China.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
No death within 30 days after surgery | 1 month after surgery for treating aortic arch disease performed
  Death from all causes would be included.
No adverse cardiovascular and cerebrovascular events within one year after surgery | 12 month after surgery for treating aortic arch disease performed
  Cerebrovascular adverse events include global neurological deficit, focal neurological deficit and spinal neurological deficit. Cardiovascular adverse events include extensive myocardial ischemia, low cardiac output syndrome, malignant arrhythmia and massive pericardial effusion.
No reoperative intervention associated with aorta occurred within one year after surgery | 12 month after surgery
  Reoperative intervention associated with aorta means unintended open or endovascular treatment of the aortic disease, excluding non-aortic surgery.

SECONDARY OUTCOMES:
Postoperative leakage | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 6 month and 12 month after surgery for treating aortic arch disease performed
  Leakage is divided into five types according to the eighth edition of Rutherford Vascular Surgery.
Patency rate of aortic arch branches | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 6 month and 12 month after surgery for treating aortic arch disease performed
  The patency of aortic arch branches (anonymous artery, left carotid artery, left subclavian artery), and whether occlusion, stenosis, thrombosis occurring in branches.
Device-related adverse events occurred | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 1 month, 6 month and 12 month after surgery for treating aortic arch disease performed
  Device-related adverse events include stent unable deploy and / or relaying to surgery, the dissection, thrombus, hematoma, pseudoaneurysm or infection of the access artery, unexplained fever continued for more than month, device-induced aortic dissection rupture or tear, displacement, infection, fracture of stent-grafts.
Postoperative new pulmonary infections | 30 days after surgery for treating aortic arch disease performed.
  New pulmonary infections occurred within 30 days after surgery.
Hypostatic pneumonia | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 1 month, 6 month and 12 month after surgery for treating aortic arch disease performed
  Long-term bed rest caused chronic congestion in the bottom of the lungs.
Lower extremity deep vein thrombosis | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 1 month, 6 month and 12 month after surgery for treating aortic arch disease performed
  It refers to the coagulation of venous blood in deep veins of the lower extremities.
Pulmonary embolism | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 1 month, 6 month and 12 month after surgery for treating aortic arch disease performed
  Endogenous or exogenous embolus clogged the main pulmonary artery or branch, causing pulmonary circulatory disorders.
Wound infection | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 1 month, 6 month and 12 month after surgery for treating aortic arch disease performed
  Wounds occurred postoperative infection.
Liver dysfunction | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 1 month, 6 month and 12 month after surgery for treating aortic arch disease performed
  Child-pugh's Grade of patient is B or C grade.
Renal dysfunction | When patient is discharged from hospital after surgery for treating aortic arch disease performed, 1 month, 6 month and 12 month after surgery for treating aortic arch disease performed
  Serum creatinine is more than 186umol/L.

OTHER OUTCOMES:
Extremities blood pressure measurement | 3 days before the surgery for treating aortic arch disease performed, 5 days after surgery for treating aortic arch disease performed
  Blood pressure of left upper limb, right upper limb, left lower limb, right lower limb

CONTACTS AND LOCATIONS:
Overall Officials: Chang Shu, Director, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (4):
- China (4):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chian-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided